CLINICAL TRIAL: NCT03558594
Title: Hypnosis and Meditation for Cancer Pain Pilot Study
Brief Title: Hypnosis and Meditation for Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rhonda Williams, PhD, Principal Investigator, VA Puget Sound Health Care System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01670
Record Dates: First submitted 2018-05-24; First posted 2018-06-15 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pain Related to Cancer; Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Hypnosis; Mindfulness

STUDY DESIGN:
Intervention Model Description: Behavioral: Self-Hypnosis Training
  Behavioral: Mindfulness Meditation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis (Experimental): Participant will have one brief meeting with a clinician in which they will learn about hypnosis and be provided with an informational booklet and with audiorecordings of hypnosis exercises. Participants will be encouraged to listen to the hypnosis recordings as much as they would like, whenever they would like to listen. The recordings are short inductions followed by therapeutic suggestions, including post-hypnotic suggestions. Participants will relax in a comfortable position with their eyes closed and will simply listen to the audio recordings that will include an induction followed by suggestions for decreased pain and improvement in co-morbid symptoms (e.g., improved mood and optimism, relaxation, sleep quality).
  Interventions: Behavioral: Hypnosis
- Mindfulness (Experimental): Participant will have one brief meeting with a clinician in which they will learn about mindfulness meditation and be provided with an informational booklet and with audio recordings of mindfulness exercises. Participants will learn Vipassana meditation by listening to audio recordings, which is the specific form of mindfulness meditation (MM) typically implemented in mindfulness research. The emphasis is placed upon developing focused attention on an object of awareness, such as the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events.Participants will be encouraged to listen to the meditation recordings as much as they would like, whenever they would like to listen.
  Interventions: Behavioral: Mindfulness
- No intervention (No Intervention): Participants will enroll in the study, but do not select a study intervention. They will complete study assessments on the same schedule as those participants who select either experimental arm.

INTERVENTIONS:
Behavioral: Hypnosis — Behavioral Condition
  Arms: Hypnosis
Behavioral: Mindfulness — Behavioral Condition
  Arms: Mindfulness

SUMMARY:
The research study involves an open label trial (i.e., participant selects one of 2 interventions) to determine whether Veterans engaged in treatment for head and/or neck cancers find either of the two available behavioral treatments for pain (Self-Hypnosis or Mindfulness) helpful in managing pain, and if the study's delivery modality (providing audio recordings and workbooks for home use) is acceptable and feasible. If neither of the 2 interventions seems appealing, the participant can participate in the study by completing the study assessments only (this option is usual care); however, the participant will not receive the study materials or one-on-one appointments with the study clinician.

DETAILED DESCRIPTION:
At any given time, 2-8 Veterans are receiving treatment for head/neck cancer at VAPSHCS, which typically involves daily appointments over a period of 6-7 weeks. Some have tumor pain prior to treatment; many of those who do not have pain at the outset experience significant pain by week 3 of treatment. Individual clinical work with these Veterans using hypnosis and mindfulness interventions has been promising.

The investigators will compare the efficacy of these two skills-based self-management approaches by looking at changes in pain and function from pre to post-treatment. This is an open label trial, so if there are sufficient participants who choose usual care, the investigators will also compare any pre-post changes to those subjects who elect usual care. Subjects will be up to 30 Veterans who are seeking treatment for head and/or neck cancer at VAPSHCS. Due to an open label model, the investigators anticipate that the treatment group size may be uneven. The investigators may find that participants select one intervention more than the others.

The investigators have designed the intervention and measures in such a way as to minimize subject burden and to limit measures to those functional outcomes relevant to this population. The investigators will emphasize implementation aspects of the evaluation, measuring feasibility, relevance, and Veteran preferences.

Knowledge generated from this study will include revealing treatment needs and preferred approaches to acute cancer pain management care for Veterans and demonstrating feasibility. The investigators anticipate that the findings will inform strategies to for making complementary meditation or self-hypnosis interventions available to Veterans dealing with cancer pain and pain related to cancer treatment. The investigators will learn if these interventions are feasible, acceptable, helpful and credible for Veterans undergoing active treatment for cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran status (defined as prior service in the US Armed Forces and eligible to receive health care services through Veterans Health Affairs)
2. 18 years of age or older
3. Undergoing head and/or neck cancer treatment at the VAPSHCS in Seattle.
4. Less than two (2) errors on the 6-item Cognitive Screener
5. Able to read, speak, and understand English

Exclusion Criteria:

1. Primary psychotic or major thought disorder as listed in participant's medical record or self-reported
2. Psychiatric or behavioral conditions in which symptoms were unstable or severe (e.g., current delirium, mania, psychosis, suicidal ideation, homicidal ideation, active substance use disorder, psychiatric hospitalization) as listed in participant's medical record or self-reported within the past six months
3. Hospitalization for psychiatric reasons involving psychosis other than suicidal ideation, homicidal ideation, and/or PTSD as noted in chart (within the past 5 years).
4. Difficulties or limitations communicating over the telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-07-28 (Estimated); Study Completion 2020-07-28 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Reported Pain Intensity from Pre to post-treatment | Baseline and 4 weeks post-baseline
  0-10 numeric scale

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Heathcare System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No